CLINICAL TRIAL: NCT06786182
Title: Effectiveness of a Pelvic Floor Contraction and Abdomino-pelvic Muscle Contraction Education Programme in Healthy Male University Students: a Pilot Study
Brief Title: Effectiveness of Abdomino-pelvic Muscle Contraction Education Programme in Healthy Male University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Marta de la Plaza, Clinical Professor, European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-442
Record Dates: First submitted 2024-10-26; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Floor; Abdominal Muscles; Abdominal Muscles/ultrasonography
Keywords: Pelvic Floor Health; Male Pelvic Floor Education; Ultrasound Imaging; Pelvic Floor Muscle Training; Physiotherapy

STUDY DESIGN:
Intervention Model Description: This study uses a randomized controlled trial (RCT) design with a parallel-group model. Participants are allocated to either a control group or an intervention group using a 1:1 ratio. The intervention group receives a structured educational program delivered via telematic resources, covering topics such as pelvic floor muscle (PFM) anatomy, function, and proper muscle activation techniques. The control group does not receive this educational intervention. Both groups undergo baseline and post-intervention ultrasound assessments to measure abdominal and PFM activation during various maneuvers, including resting, PFM contraction, the Active Straight Leg Raise (ASLR) test, and the hollowing maneuver. This model aims to evaluate the impact of the educational intervention on muscle co-contraction and activation patterns.
Who Masked: Outcomes Assessor
Masking Description: Blinding will apply to the study evaluators. The evaluators will have no knowledge about the assignment of the participants, which ensures that the evaluation of the results is unbiased and not influenced by the group to which they belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EDUCATION (Experimental): Participants receive an educational program focused on improving awareness and activation of the pelvic floor muscles and abdominal muscle synergy through telematic resources.
  Interventions: Behavioral: PFM Educational Program
- Control (No Intervention): Participants in this group receive no educational intervention and participate only in baseline and follow-up assessments of abdominal and PFM activation.

INTERVENTIONS:
Behavioral: PFM Educational Program — A structured telematic educational program covering PFM anatomy, function, and proper activation techniques. Content includes videos, visual guides, and exercises aimed at promoting PFM co-contraction and awareness.
  Arms: EDUCATION

SUMMARY:
This research study investigates the effectiveness of an educational intervention aimed at improving awareness and control of pelvic floor (PF) and abdominal muscle contractions in healthy young male university students. Using ultrasound imaging, the study measures abdominal wall muscle thickness at rest and during pelvic floor contraction, Active Straight Leg Raise (ASLR) test, and hollowing maneuvers in a randomized control trial.

DETAILED DESCRIPTION:
The study addresses the largely overlooked area of male PF health, aiming to increase awareness and improve muscle control in healthy young men. A two-group design will be used to compare abdominal and PF muscle activation between a control group and an intervention group that receives online educational content. The intervention group will participate in a telematic program covering topics such as PF anatomy, muscle function, and the importance of proper muscle activation.

The study will use diagnostic ultrasound to measure thickness changes in the transverse abdominis (TrA), internal oblique (IO), and external oblique (EO) muscles before and after the intervention in both groups under different conditions: PF rest, PF contraction, single-leg raise (ASLR) test, and the hollowing maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-30 years
* Healthy men
* Informed consent submitted, accepted and signed

Exclusion Criteria:

* Patients undergoing abdominal cavity surgery
* Patients with cognitive/proprioceptive impairments
* Patients who have had physiotherapy interventions of PFM
* Patients with low scores on the Spanish-validated SHIM sexual health questionnaire for males.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 29 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Thickness of the Transverse Abdominal Muscle (TrA) | Measured at baseline (pre-intervention) and at the end of the 4-week intervention period (post-intervention).
  Assessed at rest, during Pelvic floor (PF) contraction and during Active Straight Leg Raise (ASRL) via ultrasound,in centimetres

SECONDARY OUTCOMES:
Thickness of the External (OE) and Internal Oblique (OI) Muscles | Measured at baseline (pre-intervention) and at the end of the 4-week intervention period (post-intervention).
  Measured at rest, during PF contraction, and with the ASLR test using ultrasound, in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Angel Gonzalez de la Flor, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
No, we do not plan to share Individual Participant Data (IPD) with other researchers. We will publish aggregated results from the study, ensuring that all data is de-identified to protect participant confidentiality.

REFERENCES:
- [Background] Sapsford RR, Hodges PW, Richardson CA, Cooper DH, Markwell SJ, Jull GA. Co-activation of the abdominal and pelvic floor muscles during voluntary exercises. Neurourol Urodyn. 2001;20(1):31-42. doi: 10.1002/1520-6777(2001)20:13.0.co;2-p. PMID 11135380
- [Background] Notenboom-Nas FJM, Knol-de Vries GE, Beijer L, Tolsma Y, Slieker-Ten Hove MCP, Dekker JH, van Koeveringe GA, Blanker MH. Exploring pelvic floor muscle function in men with and without pelvic floor symptoms: A population-based study. Neurourol Urodyn. 2022 Nov;41(8):1739-1748. doi: 10.1002/nau.24996. Epub 2022 Jul 25. PMID 35876473
- [Background] Tuckett AG, Hodgkinson B, Hegney DG, Paterson J, Kralik D. Effectiveness of educational interventions to raise men's awareness of bladder and bowel health. Int J Evid Based Healthc. 2011 Jun;9(2):81-96. doi: 10.1111/j.1744-1609.2011.00208.x. PMID 21599840
- [Background] Richter LA, Gutman RE, Tefera E, Estep A, Iglesia CB. Knowledge of erectile dysfunction and pelvic floor disorders among young adults: a cross-sectional study. Can J Urol. 2015 Apr;22(2):7715-9. PMID 25891335